CLINICAL TRIAL: NCT04511013
Title: A Randomized Phase 2 Trial of Encorafenib + Binimetinib + Nivolumab vs Ipilimumab + Nivolumab in BRAF-V600 Mutant Melanoma With Brain Metastases
Brief Title: A Study to Compare the Administration of Encorafenib + Binimetinib + Nivolumab Versus Ipilimumab + Nivolumab in BRAF-V600 Mutant Melanoma With Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2000; NCI-2020-05496 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2000 (Other: SWOG); S2000 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Acral Lentiginous Melanoma; Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Cutaneous Melanoma; Metastatic Malignant Neoplasm in the Brain; Metastatic Melanoma; Metastatic Mucosal Melanoma; Pathologic Stage IV Cutaneous Melanoma AJCC v8
MeSH Terms: conditions — Melanoma; Brain Neoplasms | interventions — binimetinib; encorafenib; Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (encorafenib, binimetinib, nivolumab) (Experimental): Patients receive encorafenib PO QD on days 1-28, binimetinib PO BID on days 1-28, and nivolumab IV on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Binimetinib; Drug: Encorafenib; Biological: Nivolumab
- Arm II (nivolumab, ipilimumab) (Experimental): Patients receive nivolumab IV on day 1 of all cycles and ipilimumab IV over 30 minutes on day 1 of cycles 1-4. Cycles repeat every 21 days for 4 cycles and then every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ipilimumab; Biological: Nivolumab

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY-162; ARRY-438162; MEK162; Mektovi
  Arms: Arm I (encorafenib, binimetinib, nivolumab)
Drug: Encorafenib — Given PO
  Other Names: Braftovi; LGX 818; LGX-818; LGX818
  Arms: Arm I (encorafenib, binimetinib, nivolumab)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm II (nivolumab, ipilimumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial compares the effect of encorafenib, binimetinib, and nivolumab versus ipilimumab and nivolumab in treating patients with BRAF- V600 mutant melanoma that has spread to the brain (brain metastases). Encorafenib and binimetinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Ipilimumab and nivolumab are monoclonal antibodies that may interfere with the ability of tumor cells to grow and spread. This trial aims to find out which approach is more effective in shrinking and controlling brain metastases from melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 between participants randomized to the triplet combination of encorafenib + binimetinib + nivolumab versus the doublet combination of ipilimumab + nivolumab among participants with BRAF-V600 mutant melanoma that has metastasized to the brain.

SECONDARY OBJECTIVES:

I. To estimate the overall survival (OS) of participants in each treatment arm. II. To estimate the objective response rate (ORR) (confirmed and unconfirmed, complete and partial responses) per RECIST 1.1 in each treatment arm.

III. To estimate the intracranial response rate (ICRR), defined as confirmed and unconfirmed complete and partial response per modified RECIST for brain metastases (mRECIST).

IV. To evaluate the duration of response, per RECIST 1.1 and the duration of ICRR per mRECIST, and per Response Assessment in Neuro-Oncology (RANO)-Brain Metastases (BM) (and immunotherapy [i]RANO) in each treatment arm.

V. To evaluate the toxicity profile of each treatment arm. VI. To evaluate current and emerging radiographic response criteria (modified RECIST 1.1, modified RANO-BM and iRANO) by a retrospective blinded independent centralized review (BICR) of banked images.

BANKING OBJECTIVE:

I. To bank tumor tissue, cerebral spinal fluid (CSF), stool and blood samples for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive encorafenib orally (PO) once daily (QD) on days 1-28, binimetinib PO twice daily (BID) on days 1-28, and nivolumab intravenously (IV) on day 1. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive nivolumab IV on day 1 of all cycles and ipilimumab IV over 30 minutes on day 1 of cycles 1-4. Cycles repeat every 21 days for 4 cycles and then every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years, and then annually until 3 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically and pathologically confirmed melanoma that has metastasized to the brain
* Any primary (cutaneous, acral/mucosal, etc) or unknown origin are permitted, except that participants with uveal primary are not eligible
* Participants must have BRAF-V600 mutant melanoma documented by a Clinical Laboratory Improvement Act (CLIA)-certified laboratory
* All participants must have an magnetic resonance imaging (MRI) of the brain within 28 days prior to registration and must have central nervous system metastases with at least one measurable brain metastasis >= 0.5 cm in size (per modified RECIST 1.1) that has not been irradiated, or progressed (in the opinion of the treating physician) after prior radiation therapy. Participating sites MUST use MRI slice thickness of =< 1.5 mm and are recommended to adhere to the 'minimum' Brain Tumor Imaging Protocol for Clinical Trials in Brain Metastases (BTIP-BM) compliant MRI acquisition protocol. Computed tomography (CT) of the head cannot substitute for brain MRI. (NOTE: All central nervous system [CNS] disease must be documented on BOTH the Brain Metastases Baseline Tumor Assessment Form, using modified RECIST, and the Baseline Tumor Assessment Form [RECIST 1.1] using RECIST 1.1.)
* Participants may have measurable or non-measurable extracranial disease. All measurable disease must be assessed within 28 days prior to randomization; all non-measurable disease must be assessed within 42 days prior to randomization. Please note, while any extracranial disease will also be assessed and followed, participants are NOT required to have extracranial disease for randomization. NOTE: All disease must be assessed and documented on the Baseline Tumor Assessment Form (RECIST 1.1). CNS disease must be documented on BOTH the Brain Metastases Baseline Tumor Assessment Form, using modified RECIST, and the Baseline Tumor Assessment Form (RECIST 1.1) using RECIST 1.1
* Participants may have leptomeningeal disease
* Participants may be receiving corticosteroids for brain metastases at a dose of up to 8 mg of dexamethasone per day. The dose must not have exceeded 8 mg per day for at least 7 days prior to randomization
* Participants must have Zubrod performance status =< 2
* Participants must have complete history and physical examination within 28 days prior to randomization
* Participants must be able to swallow and retain pills
* Hemoglobin >= 8.0 g/dL (within 28 days prior to randomization)
* Absolute neutrophil count >= 1,500/mcL (within 28 days prior to randomization)
* Platelets >= 75,000/mcL (within 28 days prior to randomization)
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN) (within 28 days prior to randomization)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x institutional ULN (in participants with liver metastases =< 5 x ULN) (within 28 days prior to randomization)
* Creatinine =< 2.0 institutional ULN (within 28 days prior to randomization)
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants must be class 2B or better
* Participants with a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Participants with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 90 days prior to randomization
* Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment must have an undetectable HCV viral load prior to randomization
* Participants must agree to participate in image banking. Images must be submitted via the Triad System
* Participants must be offered the opportunity to participate in specimen and blood collections
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
* As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Exclusion Criteria:

* Participants must not have received prior systemic therapy for metastatic disease. Prior systemic therapy received only in the neoadjuvant and/or adjuvant setting (e.g., BRAF/MEK inhibitor therapy, anti-PD-1 therapy or anti-CTLA4 therapy, alfa-interferon, etc.) is permitted. If patients received prior neoadjuvant/adjuvant therapy, they must have had eventual disease relapse prior to randomization
* Participants must not have had prior radiation therapy within 7 days prior to randomization
* Participants must not be planning to require any additional form of systemic anti-tumor therapy for melanoma while on protocol treatment
* Participants must not be planning to use hormonal contraceptives
* Participants must not have a serious active infection requiring systemic therapy at time of randomization in the opinion of the treating physician
* Participants must not have active autoimmune disease that has required treatment in the past 6 months with use of biologic disease modifying agents (.e.g. infliximab, adalimumab). Patients on non-biologic disease modifying agents (e.g. methotrexate) or patients on corticosteroids =< 10 mg prednisone daily or equivalent (to treat auto-immune disease), or on replacement therapy (e.g., thyroxine, insulin) are eligible if deemed in the best interest of the patient by treating physician
* Participants must not have had grade 3 or 4 immune-related adverse events on ipilimumab or nivolumab that required more than 12 weeks of immune suppression with corticosteroids
* Participants must not have had adverse events related to encorafenib and/or binimetinib specifically, that required discontinuation of one or both drugs. (Please note this does not apply to other BRAF/MEK inhibitor drugs.)
* Participants must not be pregnant or nursing. Women/men of reproductive potential must have agreed to use an effective method of contraception. (NOTE: Patients must agree to not use hormonal contraceptives, as encorafenib can result in decreased concentration and loss of efficacy.) A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate participant chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of registration to date of first documentation of progression, or symptomatic deterioration, or death due to any cause, assessed up to 3 years after randomization
  Will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of registration to date of death due to any cause, assessed up to 3 years after randomization
  Will be assessed by Immunotherapy Response Assessment Criteria for Intracranial Metastases (RANO-BM). Will construct Kaplan-Meier plots and estimate the median OS and construct 95% Brookmeyer-Crowley Confidence intervals.
Intracranial response rate (ICRR) | Up to 3 years after randomization
  The ICRR is defined as the best response when applying modified (m)RECIST criteria. Will compare intracranial response based on assessments per mRECIST, RANO-BM and immunotherapy (i)RANO criteria based on a review of the banked images. For each of these methods, the best response to treatment will be summarized by treatment arm, the percent agreement between each pair of methods will be reported along with a 95% confidence interval, and a p-value based on a two-sided McNemar's test will be calculated.
Objective response rate | Up to 3 years after randomization
  Will be assessed by RECIST 1.1.
Duration of response | Up to 3 years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Eroglu, Principal Investigator — SWOG Cancer Research Network
Locations (331):
- United States (331):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Providence Queen of The Valley, Napa, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Sharp Memorial Hospital, San Diego, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Mercy Health - Paducah Medical Oncology and Hematology, Paducah, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - University of Michigan - Brighton Center for Specialty Care, Brighton, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Cancer Partners of Nebraska - Pine Lake, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center - 68th Street Place, Lincoln, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Wake Forest Baptist Health - Hematology Oncology - Statesville, Statesville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Columbus Oncology and Hematology Associates, Dublin, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Zangmeister Center Grove City, Grove City, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Mount Carmel New Albany Surgical Hospital, New Albany, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming